CLINICAL TRIAL: NCT03772795
Title: Changes in Pulpal Blood Flow of Teeth During Leveling and Alignment Stages of Orthodontic Treatment Using Clear Aligners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Elham Abu Alhaija, Principal Investigator - Main thesis supervisor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 262/2016
Record Dates: First submitted 2018-12-01; First posted 2018-12-11 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Alignment
Keywords: Pulpal blood flow; clear aligners; orthodontics

STUDY DESIGN:
Intervention Model Description: Two groups receiving 2 interventions. In the first group patients received fixed orthodontic appliance and in the second, they received clear aligner orthodontic appliance
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1- Alignment with fixed appliance (Active Comparator): A pre-adjusted edgewise fixed appliance (3M Gemini Uniteks, 0.022" Roth prescription brackets.Teeth alignment in this group started using round 0.014" NiTi arch wire. The 0.014" NiTi arch wire was placed into the slots of the brackets and tied with elastomers by figure of 8. During this stage, only tipping movement was applied.
  Interventions: Other: Orthodontic Alignment
- Group 2- Alignment with clear aligners (Experimental): Clear aligner orthodontic appliance (EON, Eon Dental NV, Belgium). Teeth alignment with clear aligners.
  Interventions: Other: Orthodontic Alignment

INTERVENTIONS:
Other: Orthodontic Alignment — Group 1:- Teeth alignment in this group started using round 0.014" NiTi arch wire. The 0.014" NiTi arch wire was placed into the slots of the brackets and tied with elastomers by figure of 8. During this stage, only tipping movement was applied.
  Arms: Group 1- Alignment with fixed appliance
Other: Orthodontic Alignment — Group 2: Teeth alignment using clear aligners.
  Arms: Group 2- Alignment with clear aligners

SUMMARY:
The aims of this study were to: -

* Evaluate PBF in upper and lower teeth during orthodontic alignment using fixed appliances (0.014" super elastic NiTi arch wire) at different time intervals (20min, 48h, 72h and 1 month) of initial arch wire placement.
* Evaluate the PBF in upper and lower teeth during orthodontic teeth alignment using clear aligners at different time intervals (20min ,48h, 72h and 1 month) of fitting the second aligner (first active aligner).
* Compare the PBF changes between the above two different types of orthodontic appliances (fixed appliances and the clear aligners).

DETAILED DESCRIPTION:
Aims: to evaluate the pulpal blood flow (PBF) during orthodontic teeth alignment and leveling using clear aligners (second aligner) and fixed orthodontic appliance at different time intervals of orthodontic force application.

Materials and Methods: A total of 45 subjects were subdivided in two groups: group 1: 25 subjects treated with pre-adjusted edgewise fixed appliance with 0.014 inch NiTi as the alignment arch wire and group 2: 20 subjects treated using clear aligner. In both groups, PBF was measured for the upper right and the lower left using Laser Doppler Flowmetry at different time interval (20 minutes, 48 hours, 72 hours, 1 month) after the fitting of the arch wire in group one and after the delivery of the second aligner in group two.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female subjects
* 16 or more years old
* Class I skeletal malocclusion
* mild upper and lower arches crowding. Exclusion Criteria:-
* Poor oral hygiene
* Previous orthodontic treatment
* Active periodontal disease
* Missing teeth
* Deep carious teeth
* Teeth with root resorption
* Endodontically treated teeth
* History of previous trauma
* Restoration on measured teeth
* Medical conditions affecting blood vessels
* Smoking

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Pulpal blood flow changes by the use of Laser Doppler Flowmeter (Moor lab, Moor instruments, UK) with a wavelength of 780 nm and a dental probe MP 13 (Moor instruments, UK; 2 fibers, 0.25 mm diameter, centers 0.5 mm spaced apart). | 20 minutes ,48 hours, 72 hours and 1 month
  millimeter per second

IPD SHARING:
Plan to Share IPD: Undecided